CLINICAL TRIAL: NCT00721526
Title: Disulfiram Combined With Lorazepam for Treatment of Patients With Alcohol Dependence and Primary or Secondary Anxiety Disorder
Brief Title: Disulfiram Combined With Lorazepam for Alcohol Dependence and Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michael Bogenschutz, Professor of Psychiatry, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-BOG_AA016555; K24AA016555 (NIH)
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Alcohol Dependence; Anxiety Disorder
Keywords: alcohol dependence; alcoholism; anxiety disorder; pharmacotherapy; disulfiram; lorazepam
MeSH Terms: conditions — Alcoholism; Anxiety Disorders | interventions — Disulfiram; Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Disulfiram plus lorazepam (Experimental): Disulfiram plus lorazepam
  Interventions: Drug: disulfiram plus lorazepam

INTERVENTIONS:
Drug: disulfiram plus lorazepam — Disulfiram 500mg three times weekly lorazepam 0.5-2.0 mg three times daily

SUMMARY:
The proposed design is a single-group open-label trial. Qualified consenting participants with active alcohol dependence and primary or secondary anxiety disorder will receive monitored disulfiram and lorazepam, in the context of a structured Medication Management (MM) model. In weeks 9-15 lorazepam is tapered, and disulfiram is stopped at the end of week 16. Participants who achieve 4 weeks abstinence and meet criteria for a primary anxiety disorder or mood disorder may receive ancillary medication consisting FDA-approved non-benzodiazepine treatment, with specific options for each disorder described in the protocol. Participants requiring continued treatment are referred to clinical treatment in the community at week 16, and bridging prescriptions of anxiolytic/antidepressant medication may be provided. A final follow-up assessment occurs at week 28. The primary outcomes are Percent Days Abstinent (PDA) and retention in treatment. Secondary alcohol outcomes are consequences, drinks per drinking day, remission status, and time to first heavy drinking day. Anxiety outcomes are Hamilton Anxiety Scale scores and anxiety disorder diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 and over with alcohol dependence.
* Able to provide voluntary informed consent.
* At least 4 heavy drinking days in the past 30 days.
* Primary or secondary anxiety disorder, including diagnoses of generalized anxiety disorder, panic disorder, social phobia, PTSD, obsessive-compulsive disorder, alcohol-induced anxiety disorder, or anxiety disorder not otherwise specified, ascertained by the SCID.
* Goal of abstinence.
* 2 days abstinence at the time of study entry (did not drink yesterday or today).
* Willing to come to clinic 3x/week.
* If female of child-bearing potential, willing to use approved method of contraception.

Exclusion Criteria:

* Moderate or severe withdrawal (CIWA-A greater than 15), history of withdrawal seizures or delirium tremens.
* Medical conditions (seizure disorder, sleep apnea, significantly impaired liver function, chronic or acute nephritis, symptomatic coronary artery disease, acute narrow-angle glaucoma).
* Urine drug screen positive for opioids or barbiturates.
* Hypersensitivity to thiuram derivatives.
* Pregnancy.
* Laboratory abnormalities (any LFT greater than 3 times normal, ECG evidence of ischemia, UA suggestive of nephritis, serious abnormalities of CBC).
* Need to take excluded medication (e.g. amprenavir oral solution, diazoxide oral suspension, isoniazid, lopinavir/ritonavir oral solution, metronidazole, omeprazole, phenytoins, ritonavir, tinidazole, tipranavir, warfarin, azelastine, sodium oxybate).
* Psychiatric conditions (schizophrenia, schizoaffective disorder, bipolar disorder; opioid dependence, benzodiazepine or other sedative hypnotic dependence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Bogenschutz, M. D., Principal Investigator — University of New Mexico Health Sciences Center
Locations (1):
- University of New Mexico Addiction and Substance Abuse Programs, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Disulfiram Plus Lorazepam
Started (Intent-to-treat sample) | 41
Received Study Medication | 40
Completed Week 1 Follow-up | 38
Completed Week 2 Follow-up | 37
Completed Week 4 Follow-up | 36
Completed Week 6 Follow-up | 35
Completed Week 8 Follow-up | 32
Completed Week 10 Follow-up | 29
Completed Week 12 Follow-up | 27
Completed Week 16 Follow-up (End of treatment) | 26
Completed (28 week followup) | 20
Not Completed | 21

BASELINE CHARACTERISTICS:
Arm/Group | Disulfiram Plus Lorazepam
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.66 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 20
  Hispanic | 16
  Other | 5
Region of Enrollment [Number; unit: participants]
  United States | 41
Baseline proportion abstinent days [Mean (Standard Deviation); unit: Percent] — Timeline Followback
  Percent | 0.32 (0.31)
Baseline drinks per drinking day [Mean (Standard Deviation); unit: Standard Drinks] — Timeline Followback
  Standard Drinks | 16.12 (10.97)
Baseline estimated peak blood alcohol level [Mean (Standard Deviation); unit: percent (mass/volume)] — Timeline Followback
  percent (mass/volume) | 0.34 (0.24)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Adherence
Description: Completion of 16 weeks of disulfiram treatment
Time Frame: 16 weeks
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Disulfiram Plus Lorazepam
Number analyzed (Participants) | 41
Participants | 15

2. Secondary Outcome: Percent Days Abstinent From Alcohol (Intent-to-treat Sample)
Description: As measured by Timeline Followback
Time Frame: Weeks 13-16 (Last 4 weeks of treatment)
Population: Intent-to-treat sample (Baseline value imputed for missing values)
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Disulfiram Plus Lorazepam
Number analyzed (Participants) | 41
percentage of days abstinent | 65.14 (41.004)

3. Secondary Outcome: Categorical Abstinence (Intent-to-treat Sample)
Description: As measured by timeline followback
Time Frame: Weeks 13-16 (Last 4 weeks of treatment)
Population: Percentage of 41 participants observed to be abstinent at week 16 (missing treated as non-abstinent)
Measure: Count of Participants; unit: Participants
Arm/Group | Disulfiram Plus Lorazepam
Number analyzed (Participants) | 41
Participants | 18

4. Secondary Outcome: Percent Days Abstinent From Alcohol (Among Participants Observed at Week 16)
Description: As measured by Timeline Followback
Time Frame: Weeks 13-16 (Last 4 weeks of treatment)
Population: Participants observed at week 16
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Disulfiram Plus Lorazepam
Number analyzed (Participants) | 26
Percent | 87.00 (29.569)

5. Secondary Outcome: Categorical Abstinence (Among Those Observed at Week 16)
Description: As measured by timeline followback
Time Frame: Weeks 13-16 (Last 4 weeks of treatment)
Population: observed at week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Disulfiram Plus Lorazepam
Number analyzed (Participants) | 26
Participants | 18

ADVERSE EVENTS:
Time Frame: 24 weeks following first administration of study medication
Arm/Group | Disulfiram Plus Lorazepam
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40
Other Adverse Events (participants affected / at risk) | 28/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disulfiram Plus Lorazepam (N=40)
Confusional state (Psychiatric disorders) | 1 (1) — Resulted in hospitalization, resolved without sequellae. Investigator deemed the SAE unlikely to be related to study medication or other aspects of study participation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disulfiram Plus Lorazepam (N=40)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Candida infection (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Transaminases increased (Investigations) | 3 (3)
Weight decreased (Investigations) | 1 (1)
Alcohol intolerance (Metabolism and nutrition disorders) | 12 (15) — Alcohol-disulfiram reaction
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Apathy (Psychiatric disorders) | 2 (2)
Feelings of worthlessness (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Bunion operation (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No